CLINICAL TRIAL: NCT06034782
Title: Diagnostic Accuracy of Fine Needle Aspiration in Patients With Salivary Gland Tumors,a Retrospective Study
Brief Title: Diagnostic Accuracy of Fine Needle Aspiration in Patients With Salivary Gland Tumors.
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 18/22-02-2021
Record Dates: First submitted 2022-08-19; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-08

CONDITIONS: Salivary Gland Tumor; Diagnosis
Keywords: salivary tumors; diagnostic accuracy; Fine Needle Aspiration
MeSH Terms: conditions — Salivary Gland Neoplasms; Disease | interventions — Biopsy, Fine-Needle; Histological Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with salivary gland tumors: patients with salivary gland tumors
  Interventions: Diagnostic Test: Fine Needle Aspiration; Procedure: Histologic Examination

INTERVENTIONS:
Diagnostic Test: Fine Needle Aspiration — Fine Needle Aspiration of a salivary gland tumor
  Other Names: FNA
Procedure: Histologic Examination — Histologic examination of resected salivary tumor

SUMMARY:
Tumors of the salivary glands occupy 0.5-1.2% of cases of head and neck tumors. They are primarily a surgical disease, as their treatment is basically the surgical excision. In this direction and in the context of the differential preoperative diagnosis, in addition to the imaging methods, the fine needle biopsy (FNA) was used, with which cell material is aspirated from the tumor and studied under the microscope. Although an increasing number of papers have been published in the international scientific literature over the last 5 years on the diagnostic accuracy of FNA in salivary glands, many of them are unable to quantify and omit to refer information that could affect the estimated diagnostic accuracy. Such information is for instance the clinical experience of the doctor who performs the FNA and of the one who assess the smear. The aim of this retrospective study is to evaluate the diagnostic accuracy of fine needle biopsy in adult patients with salivary gland tumor that underwent a surgical excision in two Oral and Maxillofacial Departments in Northern Greece.

The present retrospective study was carried out from 2/2021 to 4/2022 by collecting data from the files of patients who underwent surgery at the Oral and Maxillofacial Clinic of the Theageneio Cancer Hospital of Thessaloniki 1996-2022 and the General Hospital of Thessaloniki G. Papanikolaou 2015-2022. The study was conducted according to the STARD 2015 protocol.

FNA contributed significantly to the differential preoperative process in salivary gland diseases. The differential diagnosis of a lesion in benign / malignant preoperatively, with the use of FNA, enables the surgeon for a more beneficial to the patient and oncologically safer planning of the surgery. It is considered important the high sensitivity provided by the examination, as it helps to exclude with sufficient safety the possible malignancy of the tumor located in the salivary gland of the patient.

DETAILED DESCRIPTION:
This retrospective study was conducted according to the STARD 2015 protocol. A thorough retrospective analysis of patient data that were extracted from patient records of a tertiary referral hospital database was performed. The patient files which were included in the study are electronically archived at the Departments of Oral and Maxillofacial Surgery of "Theageneio Anti-Cancer Hospital of Thessaloniki" and of General Hospital of Thessaloniki "George Papanikolaou".

Patients who were included in the present study, except for clinical examination by an Oral and Maxillofacial Surgeon, also underwent at least one imaging modality (MRI, CT scan, ultrasound scan).

This retrospective study was carried out from 2/2021 to 4/2022. Data from records of patients who underwent salivary tumour surgery at the Oral and Maxillofacial Surgery departments of Theageneio Anti-Cancer Hospital of Thessaloniki 1996-2022 and of the General Hospital of Thessaloniki G. Papanikolaou 2015-2022 were collected.

The surgical treatment of all patients with salivary gland tumors who were examined by a practitioner of the two aforementioned Maxillofacial departments, was based on their chronological attendance at the outpatient clinic, while there was no attempt of grouping of them.

Based on the FNA report, FNA results were categorized as follows: Benign, Malignant, Non-diagnostic, Unavailable result. The same categories were obtained for the reference standard test, which was the histopathological examination of the resected tumor.

The sample size was calculated using the software G power analysis version 3.1.9.6. For α = 0.05 and study strength Power 0.95 a sample size of 102 patients had been obtained which was relatively smaller compared to the 128 patients that were finally included in the study.

During the data collection from the medical patient records, there were 11 (n = 11) out of 139 (n = 139) cases whose FNA result and 4 (n=4) out of 184 (n=184) whose histological result was non-diagnostic as it was not clearly concluded whether the lesion was benign or malignant. These cases were excluded from the estimation of diagnostic accuracy indicators. Likewise to the non-diagnostic results, were excluded the 145 (n = 145) FNA results that were not available.

To assess the diagnostic accuracy of FNA, a comparative process among FNA and histopathological outcomes was conducted. Sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio, ROC curve and AUC (Area Under curve) were calculated. Calculations were made using software RStudio Version 1.4.1106 © 2009-2021 RStudio, PBC "Tiger Daylily" (2389bc24, 2021-02-11) for Windows Mozilla/5.0 (Windows NT 10.0; Win64; x64) Apple Web Kit/537.36 (KHTML, like Gecko) Qt Web Engine/5.12.8 Chrome/69.0.3497.128 Safari/537.36.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years
* salivary tumor suspected
* FNA result available
* Salivary tumor surgically resected
* Histologic result available

Exclusion Criteria:

* Patients under 18 years old
* FNA result or Histologic result not available
* No tumor resection
* Other neck tumors (not salivary tumor)

Ages: 24 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with salivary tumors that examined in outpatient Oral and Maxillofacial Surgery Clinic of Anti-Cancer Hospital of Thessaloniki "Theageneio" and General Hospital of Thessaloniki "G. Papanikolaou".
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Fine Needle Aspiration in salivary tumors | Every patient underwent FNA in a time frame from 1 day to 1 month before the surgical resection of the tumor. Then, under general anesthesia the tumor was surgicaly resected and was immediately examined to the Histology Laboratory of the Hospital.
  The result FNA of salivary tumor was compared to (verified) Histologic result after tumor resection. Then Diagnostic accuracy of FNA was estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros V. Grivas, Medical, Principal Investigator — Aristotle University Thessaloniki
Locations (1):
- Aristotle University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
SN,Sex,Clinic of Origin,Date of Birth,Age, Final Result of FNA (as included in Excel database),Histological result (as included in Excel database) are available to all researchers.
Time Frame: Immediatelly available and for 6 months
Access Criteria: The excel database with the menioned individual participant data (IPD) can be available only for academical reason after email verification